CLINICAL TRIAL: NCT02029794
Title: ASPIRE Pilot: Determining Optimal Cervical Cancer Screening in a Low-resource Setting: A Randomized Controlled Trial Comparing Self-collected HPV Testing With Visual Inspection With Acetic Acid (VIA) Screening in Kampala, Uganda
Brief Title: ASPIRE Pilot: Comparing Self-collected HPV Testing With Visual Inspection With Acetic Acid Screening for Cervical Cancer
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Gina Ogilvie, Dr. Gina Ogilvie, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H13-02627
Record Dates: First submitted 2014-01-02; First posted 2014-01-08 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cervical Cancer Screening; Low Resource setting; HPV; Self-Collection; VIA
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Watchful Waiting; Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPV Self-collection (Experimental): Subjects will self-collect a cervical-vaginal sample. One time use.
  Interventions: Procedure: HPV self-colleciton
- VIA arm (Active Comparator): Standard of care in Uganda is visual inspection with acetic acid (VIA). Women randomized to this arm will undergo the following: Cervix examined by clinician using speculum and light source. Cervix then sprayed with 3-5% acetic acid, and then lesions described one minute after application of acetic acid. VIA negative no acetowhite lesions detected; positive is when dense aceto-white lesions are seen touching squamocolumnar junction
  Interventions: Procedure: visual inspection with acetic acid (VIA); Drug: 3-5% acetic acid

INTERVENTIONS:
Procedure: HPV self-colleciton — Women will self-collect a cervical sample that will be provided to an outreach worker and then labelled and sent to laboratories in Kampala for HPV testing. Women who test positive for HPV will be contacted by phone and provided with follow-up instructions.
  Other Names: Women will self-collect a cervical-vaginal specimen per instructions. Sample will then receive high-risk HPV DNA testing.
  Arms: HPV Self-collection
Procedure: visual inspection with acetic acid (VIA)
  Other Names: VIA conducted per standard of care.
  Arms: VIA arm
Drug: 3-5% acetic acid
  Arms: VIA arm

SUMMARY:
Cervical cancer remains a public health burden, particularly in developing countries such as sub-saharan Africa where the infrastructure for organized screening programs does not exist. As a result, other screening modalities (visual inspection with acetic acid) are the standard of care in such regions. It is now known, persistent infection with an oncogenic Human papillomavirus (HPV) type is a necessary precursor of cervical cancer and evidence is showing HPV testing is a potential, safe and effective alternative to cytology testing (The Pap smear). This study is evaluating the feasibility and acceptance of HPV self-collection vs. VIA in a cohort of women from Kisenyi, Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-65yrs
* Living or working in community of Kisenyi, Uganda
* Access to mobile telephone
* Fluent in Luganda, Somali or English
* Competent to provide informed consent

Exclusion Criteria:

* Known to be pregnant at study entry (self-reported)
* Complete hysterectomy
* Prior diagnosis or treatment of cervical dysplasia or cervical cancer

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06-30 (Actual); Study Completion 2015-12-29 (Actual)

PRIMARY OUTCOMES:
Histologically confirmed cervical intra-epithelial lesions grade 2 (CIN2) or greater in self-collected HPV arm and VIA arm at 12 months by colposcopy | At the 12 month follow-up visit
  Presence of low grade (CIN1) or moderate to high grade lesions (CIN2 or greater) will be compared between the two groups using chi-square testing at month 12.

SECONDARY OUTCOMES:
Uptake of HPV self-collection compared to VIA in women in Kampala, Uganda | One Year
  Proportion of women who provide HPV self collected specimen or who attend initial VIA will be compared between groups using Pearson's Chi-square test. Proportion of women who complete all recommended follow-up assessments and treatment (if required) will be compared between groups using chi-square testing.
Prevalence rates of high-risk HPV in the self-collection arm. | One year
Assess screen positive rates by nurse-midwife exam in VIA arm | One year
Evaluation of adverse events or complications documented at time of sample collection, 4-6 weeks after cryotherapy and at 12 and 36 months by study questionnaire | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Gina Ogilvie, MD FCFP DrPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada